CLINICAL TRIAL: NCT05260203
Title: Evaluation of Performance and Safety of APP RITA in Increasing the Therapeutic Adherence of Onco-Hematological Patients - a Prospective Monocentric Pre-Market Study with a Historical Group of Comparison
Brief Title: MargheRITA (Remote Intelligence for Therapeutic Adherence)
Acronym: MargheRITA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advice Pharma Group srl (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CO-09-A02
Record Dates: First submitted 2021-12-30; First posted 2022-03-02 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2023-02

CONDITIONS: Multiple Myeloma; Solitary Plasmacytoma; Amyloidosis; Chronic Myeloid Leukemia; Chronic Lymphocytic Leukemia; T Cell Non-Hodgkin Lymphoma; Lymphocytic Lymphoma; Hodgkin Lymphoma; B-cell Non Hodgkin Lymphoma; Acute Myeloid Leukemia; Myelodysplasia; Chronic Myeloproliferative Disorder; Treatment Adherence; Treatment Adherence and Compliance
Keywords: Digital Therapeutics; Digital Medicine; Oncologic treatment; Hematologic treatment; Adherence; Software; Software Medical Device; Quality of life; Digital Therapy
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Amyloidosis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, T-Cell; Hodgkin Disease; Lymphoma, B-Cell; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts; Myeloproliferative Disorders; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: This is a prospective, interventional, confirmatory investigation, pre-market study, with a historical group of comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- App RITA (Experimental): The interventional study group will use the Device Rita, an application that allow the oncological and onco-hematological patients to receive and communicate information about the quality of life and about the treatment related adverse events, providing a support in the therapy management. The access to the app functionalities is granted when the physician habilitates the personal profile. The app can be also used from people designated from the patient as caregiver, who can view the data inserted by the patient and, if enabled, they can insert the data for the patient.
  Interventions: Device: RITA (App)
- Retrospective Historical (No Intervention): This clinical trial has no control intervention; on the other hand, the clinical outcomes of this treatment will be compared with the retrospective clinical data obtained from a historical group of comparison. The historic control used in this clinical trial is specifically selected to reflect the endpoints. According to a feasibility phase of this study, the information on the date of start and end of treatments is routinely collected in the medical records of patients, and for this reason, these data are potentially already available for the historical control group.

INTERVENTIONS:
Device: RITA (App) — The RITA "Remote Intelligence for Therapeutic Adherence" application was designed, on the doctor's side, as a support for the management of the onco-hematological patient and, on the patient's side, as a first aid tool for the management of the most common problems, as well as an efficient and "non-invasive" means of communication with the doctor. The system also allows the caregiver and general practitioner to be included in the communication group.
  The added value of the app consists in improving the relationship between the patient and the doctor, creating an effective communication channel, increasing the safety the patient has when facing his difficult path, reducing the number of visits to the facility and, in general, making those visits more efficient, thus creating savings both in terms of time and resources.
  Arms: App RITA

SUMMARY:
It is essential to improve clinical efficiency and management of hematological and oncological patients treated on an outpatient basis. The most promising operative way to achieve this result is the development of tele-oncology platforms, that allow not only a telemedicine visit, but also the patient support in the daily management of the disease and related disorders, as well as treatments and their complications. In this perspective, the RITA communication platform should be able to support the patient, the caregiver, the physician and the general practitioner in the management of the disease and its treatments.

DETAILED DESCRIPTION:
Summary description of the investigational device:

The RITA "Remote Intelligence for Therapeutic Adherence" application was designed, on the doctor's side, as a support for the management of the onco-hematological patient and, on the patient's side, as a first aid tool for the management of the most common problems, as well as an efficient and "non-invasive" means of communication with the doctor. The system also allows the caregiver and general practitioner to be included in the communication group.

The added value of the app consists in improving the relationship between the patient and the doctor, creating an effective communication channel, increasing the safety the patient has when facing his difficult path, reducing the number of visits to the facility and, in general, making those visits more efficient, thus creating savings both in terms of time and resources. RITA is also designed to communicate and receive information on the quality of life and side effects, thus making the medical doctor aware of the progress of treatments in his patient population.

Often occurs that the mild drug/disease related symptoms that the patient perceive during the treatment period are underestimated, leading to a more severe symptomatology that could impair the patient adherence to treatment. Thanks to the app RITA, on the patients side it will be easier to notify their daily physical condition, while on the physician side it will be easier to manage and solve the mild symptoms the patient could face during the treatment period, improving the overall adherence to the treatment.

The mobile app, which can also be used on a conventional desktop or laptop, aims to optimize the interaction between the onco-hematological patient and the referring physician. The hospital doctor will have access to the website, in order to manage all the functions through the appropriate dashboard.

Intended purpose of the investigational device in the proposed clinical investigation:

The application allows, on the patient side, to:

* record the relevant symptoms, with a simple classification, to be reported to the doctor at the next visit;
* record Quality of Life (QoL) data at pre-selected timepoints;
* inform the doctor about the necessary drug prescriptions;
* contact the doctor for advice for the same day;
* receive suggestions, through both video and text, specific to the most common problems that patients may face (the advice can be specific in relation to the type of treatment carried out). The consultation is personalized by the attending physician based on the clinical characteristics of the patient, and the personalization takes place through the selection of a series of profiles created for the different types of patients (e.g. fever in patients with mild, moderate or severe impaired immune system, etc.);
* monitor relevant clinical parameters, such as: temperature, heart rate, blood pressure, oxygen saturation, respiratory rate, glycemia;
* report information on the quality of life by filling in a specific questionnaire at defined timepoints;
* monitor the intake of specific drugs;
* manage contacts with the caregiver.

While, on the hospital doctor side, the website allows to:

* have a quick and complete overview of the problems suffered by the patient in the period since the last visit, thus making the visit faster and more productive;
* have information related to different and relevant clinical parameters measured and inserted from the patient, including temperature, heart rate, blood pressure, oxygen saturation, respiratory rate, glycemia; the collection of this information will allow the doctor to have patient's information necessary to carry out the appropriate clinical assessments on response to therapy, stability and/or relapse of the disease. For example, the temperature value can be communicated directly to the doctor to anticipate the prescription of the antibiotic;
* facilitate the home management of the most common clinical problems that the patient can face, through videos and texts, customizable by the doctor, which explain how to deal with the most common symptoms in an initial phase;
* know in advance the drug prescriptions needed by the patient, thus allowing to assign the prescription activity to the support staff;
* collect in a single "container" all daily communications of patients, which are normally dispersed in a multiplicity of channels (telephone calls, faxes, e-mails), in order to be able to manage them conveniently;
* easily communicate with the caregiver;
* monitor patients' QoL prospectively.

Description of the specific medical procedures involved in the use of the investigational device:

Possible features of the RITA app:

* possibility of reminder for drugs intake;
* possibility of creating a grading or threshold levels in case of symptoms such as fever (e.g., temperature at 37.1°C or 39°C); then a response is generated based on the grading (e.g., "go to the emergency room" or "take a drug'');
* possibility for the doctor to select the advice to send to the patient;
* possibility for the doctor to select the type of pathology and the characteristics of the patient (e.g., immunodepressed patient);
* possibility of integrating diets and ad hoc menus based on drugs administered;
* possibility of inserting tutorials (e.g., how to send blood counts values);
* possibility of uploading contents: both the doctor and the patient can send texts or multimedia contents;
* possibility of sending a warning about adherence to therapy both to the doctor and to the caregiver.

Rationale for benefit-risk ratio.

The major risk for onco-hematologic patients is the progression of their underlying disease and the consequent reduction in the quality of life, which can be accelerated by a reduced adherence to the therapy. Risks associated with participation in the clinical investigation are the same as the risks identified for the general use. No additional risk is identified, specifically related to the participation in the clinical investigation, as the patient does not receive a lowered standard of care. Moreover, no special risks are reported due to the use of applications for adherence to treatment.

Therefore, the potential risks identified in association with the treatment administered with the App RITA are justified by the anticipated benefits resulting from the implementation of the standard of care aiming at improving the patients' involvement in their own health management and intended increase of adherence to treatment.

Primary Objective

The primary objective is the evaluation of patients' compliance to treatment through the use of the app RITA, thanks to more efficient management of the patients' mild symptoms that could, if not promptly treated, lead to a more severe condition and sometimes to the treatment interruption.

Secondary Objectives

* Reduction of grade 3-4 treatment-related adverse events.
* Reduction in the number of visits to the emergency room for complications not requiring hospitalization: careful monitoring of the patient, both during follow-up visits and through the use of the RITA app, allows for better control of complications, reducing the patient's need to access the emergency room.
* Reduction in the number of visits to the emergency room for severe complications requiring hospitalization: careful monitoring of the patient, both during follow-up visits and through the use of the RITA app, allows for better control of complications, reducing the patient's need to access the emergency room.
* Reduction in the average number of days in hospital stay: through careful monitoring of the patient, both during follow-up visits and through the use of the RITA app, it is possible to reduce the occurrence of severe complications that may require the patient to be hospitalized. This objective evaluates the average number of days of hospitalization of the patient due to the onset of complications.
* Improvement in the quality of life perceived by the patient: the use of tools in order to assess the quality of life (for example: questionnaires) allows the medical doctor to check the patient's perception of health and identify any limitations in daily life activities. A constant survey allows to identify timely and more effective solutions aimed at improving the patient's quality of life.
* User Experience: the use of digital tools (for example: apps, web systems, etc..), to support the doctor-patient clinical health interactions, allows continuous monitoring of the patient both with respect to any clinical complications and with regard to a worsening of the quality of life. The indicator monitors the overall degree of patient satisfaction in relation to the use of the RITA app. In this way, it is possible to verify the real effectiveness of the app and intercept any elements of attention with respect to the features present.

Primary Endpoint The primary endpoint is the evaluation of the therapeutic adherence measured as at least the 80% of the relative dose intensity (defined as the ratio of delivered dose intensity to the prescribed referenced dose intensity, expressed as a percentage) during the study period. The effectiveness of the RITA app use will be evaluated by comparing results on therapeutic adherence with a historical group of cancer patients.

Secondary Endpoint

Secondary endpoints based on the comparisons between groups:

* Number of visits to the emergency room for complications not requiring hospitalization: analysis will be performed on the population enrolled in the trial versus an historical control, evaluating the recorded number of visits to the emergency room for minor complications not requiring hospitalization. This information will be obtained by consulting the management control of the hospital or the emergency room system.
* Number of visits to the emergency room for severe complications requiring hospitalization: analysis will be performed on the population enrolled in the trial versus an historical control, evaluating the recorded number of visits to the emergency room for severe complications requiring hospitalization. This information will be obtained by consulting the management control of the hospital or the emergency room system.
* Average number of days in hospital stay: analysis will be performed on the population enrolled in the trial versus an historical control, dividing the number of days in hospital stay for hematological patients by the number of hematological patients taken care of. This information will be obtained by consulting the management control of the hospital.
* Number of AE/minor complications not requiring assistance notified by the patient during the study period, through the app RITA and directly during the clinical visit, compared to the historical control group.
* To measure quantitatively the therapeutic adherence through the mean relative dose intensity (defined as the ratio of delivered dose intensity to the prescribed referenced dose intensity, expressed as a percentage) during the study period.

Secondary endpoints on the safety assessment of RITA APP:

* Occurrence of individual adverse events (%) reported during the follow-up period, during the user session, and during intervals between one use session and the following.
* Occurrence of device adverse events (%) during the user session.

Medical Device CLASS IIA

Determination of Sample Size With a total of 112 patients (56 patients in the interventional arm and 56 in the patient-level historical group), this investigation will have 80% power to detect a 20% improvement in treatment adherence (i.e., in the intervention group, 90% or more as compared to 70%) (Passardi et al., 2022), with a one-sided type I error rate of 0.05. We set a goal of enrolling 124 patients to account for a drop-out rate of 10% (Passardi et al., 2022), with a consequent enrollment of 62 patients per arm.

Statistical Analyses

In the primary analysis, all the patients observed until the end of the study will be included.

Patients in the historical group will be matched with patients in the prospective interventional study according to cancer diagnosis and type of anticancer treatment.

The main characteristics of the patients will be reported using descriptive analyses by tabulating frequencies and percentages (categorical variables) and mean and median values, standard deviations (SD), quartiles and extreme values (continuous variables). With reference to comparison between groups, odds ratios (OR) and 95% confidence intervals (CI) will be calculated to evaluate the effectiveness of the RITA app, using logistic regression models. The statistical significance limit will be accepted as 5%, and the results below this value (P < .05) will be considered statistically significant. Comparisons within group (i.e., in the interventional study group) will be performed by using the paired t-test or the corresponding Wilcoxon signed-rank test, a non-parametric test for paired samples, after checking data were normally distributed (based on the Shapiro-Wilk statistic). Comparisons between groups (i.e., interventional and historical) for continuous data will be analysed using a two-sided Student's t-test, after checking data were normally distributed (based on the Shapiro-Wilk statistic) and a two-sided Wilcoxon's rank-sum test otherwise. For categorical data comparisons between groups will be performed by using the contingency table analysis with the Chi-square or Fisher's exact test, when appropriate. Explorative analyses, with descriptive purpose only, will be performed in the subgroups of potential determinants of adherence of anticancer treatments, including age, gender, educational status, stage of disease, comorbidities, poly-pharmacy and complexity of oral anticancer regimens(weekly/daily). Adverse events occurring during the study follow-up will be tabulated.

QUALITY ASSURANCE AND CONTROL

All participant data relating to the study will be recorded on eCRF. The investigator is responsible for verifying that data entries are accurate and correct by electronically signing the eCRF.

The investigator must maintain accurate documentation (source data) that supports the information entered in the eCRF.

The investigator must permit study-related monitoring, audits, IRB/IEC review, and regulatory agency inspections and provide direct access to source data documents.

Monitoring details describing strategy (eg, risk-based initiatives in operations and quality such as Risk Management and Mitigation Strategies and Analytical Risk-Based Monitoring), methods, responsibilities, and requirements, including handling of noncompliance issues and monitoring techniques (central, remote, or on-site monitoring) are provided in the monitoring plan.

The sponsor or designee is responsible for the data management of this study including quality checking of the data.

The sponsor assumes accountability for actions delegated to other individuals (eg, Contract Research Organizations).

Study monitors will perform ongoing source data verification to confirm that data entered into the eCRF by authorised site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP, and all applicable regulatory requirements.

Data Management System The CRFs in this trial are implemented electronically using a dedicated EDC system (ICE, Integrated Clinical Trial Environment, Advice Pharma) that fulfils the legal requirements for clinical trials. The EDC system is activated for the user only after successfully passing a formal test procedure. All data entered in the EDC are stored on a Linux server in a dedicated Oracle database.

Monitoring The study will be monitored on a regular basis by the Sponsor's adequately qualified and trained clinical Monitors throughout the study period to ensure the proper conduct of the clinical Investigation.

The purposes of study monitoring are to verify that the rights and well-being of study subjects are protected, that the reported study data are accurate, complete and verifiable against the source documents, and that the study is conducted in accordance with the current clinical investigation plan, Good Clinical Practice guideline (UNI EN ISO 14155) and applicable regulatory requirements.

Audits and Inspections Upon request by the Sponsor, on-site study audits may be conducted in order to ensure the study is in compliance with GCP, applicable regulatory requirements, and the clinical investigation plan. The auditing activities may also be conducted after study completion.

ELIGIBILITY:
Inclusion Criteria:

* Patients who understand and voluntarily sign an informed consent form (ICF) prior to any study related procedures being conducted;
* Patients who are ≥ 18 years old;
* Patients who are diagnosed with a onco-hematologic disease, namely: Symptomatic Multiple Myeloma, Solitary Plasmocytoma, Amyloidosis, Chronic Myeloid Leukemia, Chronic Lymphocytic Leukemia, Lymphocytic Lymphoma, Hodgkin Lymphoma, B cells non-Hodgkin Lymphoma, T cells non-Hodgkin Lymphoma, Acute myeloid Leukemia, Myelodysplasia, Chronic Myeloproliferative Disorder;
* Patients who receive a standard of care therapy for their disease, independently from the route of administration;
* Patients in their first or subsequent line of therapy;
* Patients at the beginning of the treatment, or during therapy;
* Life expectancy > 6 months.

Exclusion Criteria:

* Patients treated with radiotherapy only;
* Presence of clinical conditions that will impair the adherence to the treatment (ie, concomitant tumor on treatment, severe neurologic disease, drug or alcohol abuse etc.);
* Patient unable to use a smartphone and/or a computer (ie blindness, inability to use a smartphone or a computer etc.);
* Major psychopathology or cognitive impairment likely in the judgment of the research staff to interfere with the participation or completion of the protocol;
* Patient enrolled in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2022-06-04 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Evaluating changes in actual dose intensity | Daily/ Assessment at each month for three months
  The primary outcome is defined as the comparison between the proportion of patients with at least 20% of increase in the relative dose intensity (defined as the ratio of delivered dose intensity to the prescribed referenced dose intensity, expressed as a percentage) of anticancer treatment during the study period in the two arms (i.e., intervention and historical group). The actual delivered dose intensity will be evaluated at each follow up visit through the drug accountability performed onsite.

SECONDARY OUTCOMES:
Number of grade 3-4 adverse events | Daily/ Assessment at each month for three months
  Incidence of grade 3-4 treatment-related adverse events
Number of visits to the Emergency Room | Daily/ Assessment at each month for three months
  Number of visits to the emergency room for complications not requiring hospitalization Number of visits to the emergency room for severe complications requiring hospitalization
Number of days in hospital | Daily/ Assessment at each month for three months
  Average number of days in hospital stay
Quality of life change - Questionnaire EQ-5D-5L | Daily/ Assessment at each month for three months
  Evaluation of changes in the quality of life perceived by the patients using the validated questionnaire for data collection EQ-5D-5L
Quality of life change - Questionnaire EORTC QLQC30 | Daily/ Assessment at each month for three months
  Evaluation of changes in the quality of life perceived by the cancer patients using the validated questionnaire for data collection EORTC QLQC30
RITA APP Experience evaluation | Daily/ Assessment at each month for three months
  User Experience in using the RITA APP, through the questions proposed by the app about the user satisfaction

OTHER OUTCOMES:
Minor complications | Daily/ Assessment at each month for three months
  Number of AE/minor complications not requiring assistance notified by the patient during the study period, through the app RITA and directly during the clinical visit, compared to the historical control group
Safety Outcome - Adverse events | Daily/ Assessment at each month for three months
  Occurrence of individual adverse events (%) reported during the follow up period, during the use session, and during intervals between one use session and the following Occurrence of device adverse events (%) during the use session

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Flavio Ferri, Study Director — Advice Pharma Group S.r.l.
Locations (1):
- ASST Santi Paolo e Carlo - SSD Ematologia - Neoplasie Ematologiche P.O. San Carlo, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sandstrom M, Wilen J, Oftedal G, Hansson Mild K. Mobile phone use and subjective symptoms. Comparison of symptoms experienced by users of analogue and digital mobile phones. Occup Med (Lond). 2001 Feb;51(1):25-35. doi: 10.1093/occmed/51.1.25. PMID 11235824
- [Background] Oftedal G, Wilen J, Sandstrom M, Mild KH. Symptoms experienced in connection with mobile phone use. Occup Med (Lond). 2000 May;50(4):237-45. doi: 10.1093/occmed/50.4.237. PMID 10912374
- [Background] Chia SE, Chia HP, Tan JS. Prevalence of headache among handheld cellular telephone users in Singapore: a community study. Environ Health Perspect. 2000 Nov;108(11):1059-62. doi: 10.1289/ehp.001081059. PMID 11102297
- [Background] Koivisto M, Haarala C, Krause CM, Revonsuo A, Laine M, Hamalainen H. GSM phone signal does not produce subjective symptoms. Bioelectromagnetics. 2001 Apr;22(3):212-5. doi: 10.1002/bem.41. PMID 11255218
- [Background] Hocking B. Preliminary report: symptoms associated with mobile phone use. Occup Med (Lond). 1998 Sep;48(6):357-60. doi: 10.1093/occmed/48.6.357. PMID 10024730
- [Background] Hietanen M, Hamalainen AM, Husman T. Hypersensitivity symptoms associated with exposure to cellular telephones: no causal link. Bioelectromagnetics. 2002 May;23(4):264-70. doi: 10.1002/bem.10016. PMID 11948605
- [Background] Wilen J, Sandstrom M, Hansson Mild K. Subjective symptoms among mobile phone users--a consequence of absorption of radiofrequency fields? Bioelectromagnetics. 2003 Apr;24(3):152-9. doi: 10.1002/bem.10101. PMID 12669297
- [Background] Koivisto M, Revonsuo A, Krause C, Haarala C, Sillanmaki L, Laine M, Hamalainen H. Effects of 902 MHz electromagnetic field emitted by cellular telephones on response times in humans. Neuroreport. 2000 Feb 7;11(2):413-5. doi: 10.1097/00001756-200002070-00038. PMID 10674497
- [Background] Oftedal G, Straume A, Johnsson A, Stovner LJ. Mobile phone headache: a double blind, sham-controlled provocation study. Cephalalgia. 2007 May;27(5):447-55. doi: 10.1111/j.1468-2982.2007.01336.x. Epub 2007 Mar 14. PMID 17359515
- [Background] Rubin GJ, Hahn G, Everitt BS, Cleare AJ, Wessely S. Are some people sensitive to mobile phone signals? Within participants double blind randomised provocation study. BMJ. 2006 Apr 15;332(7546):886-91. doi: 10.1136/bmj.38765.519850.55. Epub 2006 Mar 6. PMID 16520326